CLINICAL TRIAL: NCT02827357
Title: Review of Responses to Systemic Chemotherapy of Patients With Non-small Cell Lung Cancer Harboring a Known Somatic Activating HER2 Mutation
Brief Title: Responses to Chemotherapy of Patients With Non-small Cell Lung Cancer Harboring a Known Somatic Activating HER2 Mutation
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 14 7305 03
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No specific intervention — Clinical, drug and data collection : characteristics of patients (age, sex and histology), non HER 2-directed treatments including response and duration of response

SUMMARY:
This chart review describe the response to systemic chemotherapy of patients with non-small cell lung cancer (NSCLC) harbouring a known somatic activating human epidermal growth factor receptor 2 (HER2) mutation. The analysis of this data will provide an initial description of the response to systemic chemotherapy in patients with NSCLC harboring an activating HER2 mutation in order to inform the design and powering of future randomized controlled clinical trials of HER2-directed therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients with advanced nonsmall-cell lung cancer
* known HER2 exon-20 insertion
* treated with chemotherapy and/or HER2-targeted drugs

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with advanced nonsmall-cell lung cancer (NSCLC), a known HER2 exon-20 insertion, treated with chemotherapy and/or HER2-targeted drugs
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall response rate | 24 months

SECONDARY OUTCOMES:
Median progression-free survival (PFS) with conventional chemotherapy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: MAZIERES Julien, MD PhD, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No